CLINICAL TRIAL: NCT00731263
Title: A Phase I/II, Open-Label, Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the Tor Kinase Inhibitor AZD8055 Administered Orally to Patients With Advanced Solid Tumours.
Brief Title: A Study of Tor Kinase Inhibitor in Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1600C00001; 2008-002606-19
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
Keywords: Cancer; Advance solid tumours; Dose Escalation; Preliminary efficacy; AZD8055; Tor kinase inhibitor; Oral administration
MeSH Terms: conditions — Neoplasms | interventions — (5-(2,4-bis((3S)-3-methylmorpholin-4-yl)pyrido(2,3-d)pyrimidin-7-yl)-2-methoxyphenyl)methanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The study will start with AZD8055 formulated in a liquid solution prior to the tablet formulation becoming available. The tablet formulation will be introduced in Part A at the beginning of a new cohort at an appropriate dose, no higher than the dose of the liquid formulation in the last completed evaluated cohort. Oral solution or tablet, single dose on Day 1 Part A, twice daily ascending dosing from day 8 onwards (until maximum tolerated dose is reached), cycles of 28 days treatment.
  Interventions: Drug: AZD8055

INTERVENTIONS:
Drug: AZD8055 — Oral solution or tablet, single dose on Day 1 Part A, twice daily ascending dosing from day 8 onwards (until maximum tolerated dose is reached), cycles of 28 days treatment.

SUMMARY:
The purpose of the study is to assess the safety, tolerability and pharmacokinetics of AZD8055 and determine the maximum tolerated dose to take into phase II trials.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of an advanced solid malignant tumour (or lymphoma Part A only)
* Cancer which is refractory to standard therapies or for which no standard therapy exists, patients with measurable or non-measurable disease (according to RECIST criteria) can be recruited to Part A
* Evidence of post-menopausal status or negative urine/serum pregnancy test for pre-menopausal female patients

Exclusion Criteria:

* Patients with severe laboratory abnormalities for haematology, liver or renal function. Also treatment with any haemopoietic growth factors are not allowed within two weeks from first dose of study drug.
* Patients with abnormal fasting glucose, have type I or II Diabetes or have uncontrolled blood fats and cholesterol
* Patients with a history of neurological disease, peripheral or central neuropathy, brain metastases or family history of myopathy are excluded
* Patients with severe cardiac condition of ischemia, impaired ventricular function and arrhythmias, evidence of severe or uncontrolled systemic or current unstable or uncompensated respiratory or cardiac conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD8055 | Assessed at all visits

SECONDARY OUTCOMES:
To identify early signals of anti-tumour activity | Visits 1, 5, and 9 and 11
To identify early signals of anti-tumor activity | Visits 1, 5, 9 and 13

CONTACTS AND LOCATIONS:
Overall Officials: Prof Stan Kaye, Principal Investigator — Royal Marsden Hospital, Sutton, Surrey, England, SM2 5PT; Dr Carol Aghajanian, Principal Investigator — Memorial Sloan-Kettering Cancer Centre, 1275 York Avenue, New York, NY 10065, USA; Dr Aung Naing, Principal Investigator — MD Anderson Cancer Centre, 1515 Holcombe Blvd, Houston, Texas, USA; Professor Eric Raymond, Principal Investigator — Hôpital Beaujon, 100, Boulevard du Général Leclerc, 92118 Clichy Cedex, France
Locations (4):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Research Site, Clichy, France
- Research Site, Sutton, Surrey, United Kingdom